CLINICAL TRIAL: NCT03408691
Title: The Effect of a Probiotic Strain on Stress-related Intestinal Hyperpermeability in Adult Humans.
Brief Title: PRObiotic and Stress-related PERmeability
Acronym: ProSPer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S60969
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2018-01

CONDITIONS: Permeability; Increased
Keywords: probiotic; permeability; stress

STUDY DESIGN:
Intervention Model Description: Single-site exploratory randomized, controlled interventional trial with a parallel group design: double blind with Test and Control arm + open label arm without intervention.
Who Masked: Participant, Investigator
Masking Description: double blind only in Test and Control arm open label in arm without intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test product (Active Comparator): Fresh fermented dairy drink containing probiotic strain consumed as follows: one bottle (100g) BID for 6 weeks
  Interventions: Dietary Supplement: Fresh fermented dairy drink containing probiotic strain
- Control product (Placebo Comparator): Acidified dairy drink without ferment consumed as follows: one bottle (100g) BID for 6 weeks
  Interventions: Other: Acidified dairy drink without ferment
- No product (No Intervention): no product

INTERVENTIONS:
Dietary Supplement: Fresh fermented dairy drink containing probiotic strain — Fresh fermented dairy drink containing probiotic strain consumed as follows: one bottle (100g) BID for 6 weeks.
  Arms: Test product
Other: Acidified dairy drink without ferment — Acidified dairy drink without ferment consumed as follows: one bottle (100g) BID for 6 weeks.
  Arms: Control product

SUMMARY:
This is a single-site exploratory study aiming to demonstrate the effect of a fresh fermented dairy drink containing a probiotic strain on stress-related intestinal hyperpermeability in students defending a bachelor's or master's thesis in front of a jury at the University of Leuven (Belgium).

DETAILED DESCRIPTION:
The study is conceived as a single-site exploratory study with a randomized, controlled, parallel group design. There will be a double blind with 2 intervention arms (Test product with probiotic and acidified milk Control) plus an extra open label arm without intervention in a 2:2:1 ratio. The goal of the open-label arm is to confirm our previous data on the effect of stress on small intestinal permeability (see reference), without powering the study to detect a significant difference within this open-label arm. The participants and the investigators are blinded to the allocation to the probiotic vs. acidified milk control arm. However, there is no blinding in the arm without intervention.

In vivo intestinal permeability and salivary markers of psychological stress and activation of the autonomous nervous system will be measured and questionnaires will be completed at 4 different test days: baseline (V2), two weeks after randomization (V3), during an oral defense of a master's or bachelor's thesis (V4) and finally after pretreatment with Indomethacin (V5).

The 5 study visits are organized around the thesis defence (D0):

V1 (screening + inclusion) takes place within 2 to 3 weeks prior to the randomization.

V2 (baseline + randomization) will take place between D-35 to D-27. V3 (randomization + 2 weeks) will take place at D-14 +/-1day. V4 (thesis defense) is D0 and organized by the University. V5 (Indomethacin) will take place at D+14 +/-1day.

For subjects in the intervention arm (Test product with probiotic and acidified milk Control), products will be supplied (for 1 week). In addition, alternate product supply will take place at D-21, D-7 and D+7 (each one +/-1day).

ELIGIBILITY:
Inclusion Criteria:

* Student defending a bachelor's or master's thesis in front of a jury
* Age 20 till 30 years (both included), both genders
* Subject, upon briefing of the content of the present study, fully understanding and agreeing to its objective and having given written (dated and signed) informed consent form to take part in the study
* Subject willing to consume 2 units of investigational product per day during the investigational product consumption period.
* For females: If of child bearing potential, female subjects must be using or complying with methods of contraception
* Subject willing to strictly follow dietary/medication instructions for the entire duration of the study
* Subject must have access to a refrigerator with adequate space to store the investigational products according to the labels' storage recommendations and a freezer for the cooling elements in the transport bag

Exclusion Criteria:

* Subject with chronic gastrointestinal disorders or symptoms, type 1 or type 2 diabetes mellitus, psychiatric disease including but not limited to depression (screened by PHQ-9) and general anxiety disorder (screened by GAD-7), celiac disease, food allergy or a history of atopic conditions (eczema, allergic asthma, allergic rhinoconjunctivitis) requiring active treatment
* Subject with allergy or intolerance to non-steroidal anti-inflammatory drugs (NSAID)
* Subject with first degree relatives with coeliac disease, inflammatory bowel disease (IBD) or type 1 diabetes
* Subject with known or suspected lactose intolerance or suspected allergy or hypersensitivity to any component of the study product(s) (e.g. milk protein)
* Subject receiving (currently or in the 2 last weeks) systemic treatment or topical treatment likely to interfere with evaluation of the study parameters: antibiotics, intestinal or respiratory antiseptics, anti-rheumatics, NSAIDs and steroids prescribed in chronic inflammatory diseases.
* Active smoker with at least 7 cigarettes per week
* Subject consuming regularly (>1/week) more than 3 units of alcohol per day.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Lactulose-Mannitol Ratio (LMR) during the stress condition vs. baseline | oral administration of Test or Control product for 4 weeks before stress condition
  LMR or in vivo small intestinal permeability during stress condition vs. baseline in the Test product with probiotic compared to the acidified milk Control arm

SECONDARY OUTCOMES:
LMR during administration of Test or Control product vs. baseline | oral administration of Test or Control product for 2 weeks
  LMR or in vivo small intestinal permeability during administration vs. baseline within each intervention arm and between groups.
LMR after indomethacin vs. baseline | oral administration of Test or Control product for 6 weeks before indomethacin
  LMR or in vivo small intestinal permeability after indomethacin vs. baseline within each intervention arm and between groups
Salivary cortisol during the stress condition vs. baseline | oral administration of Test or Control product for 4 weeks before stress condition
  Salivary cortisol during the stress condition vs. baseline within each intervention arm and between groups
Subjective anxiety levels (STAI state) during the stress condition vs. baseline | oral administration of Test or Control product for 4 weeks before stress condition
  Subjective anxiety levels (STAI state) during the stress condition vs. baseline within each intervention arm and between groups

CONTACTS AND LOCATIONS:
Overall Officials: Tim Vanuytsel, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgie, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanuytsel T, van Wanrooy S, Vanheel H, Vanormelingen C, Verschueren S, Houben E, Salim Rasoel S, Tomicronth J, Holvoet L, Farre R, Van Oudenhove L, Boeckxstaens G, Verbeke K, Tack J. Psychological stress and corticotropin-releasing hormone increase intestinal permeability in humans by a mast cell-dependent mechanism. Gut. 2014 Aug;63(8):1293-9. doi: 10.1136/gutjnl-2013-305690. Epub 2013 Oct 23. PMID 24153250
- [Derived] Wauters L, Van Oudenhove L, Accarie A, Geboers K, Geysen H, Toth J, Luypaerts A, Verbeke K, Smokvina T, Raes J, Tack J, Vanuytsel T. Lactobacillus rhamnosus CNCM I-3690 decreases subjective academic stress in healthy adults: a randomized placebo-controlled trial. Gut Microbes. 2022 Jan-Dec;14(1):2031695. doi: 10.1080/19490976.2022.2031695. PMID 35130109